CLINICAL TRIAL: NCT05803668
Title: Incidence of Cholelithiasis After Bariatric Surgery in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Mohamed, Resident of general surgery of sohag university hospital, Sohag University
Other Study IDs: soh-Med-23-03-06MS
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who developed gall stones
- patients who did not develope gall stones

SUMMARY:
To study the incidence and predictors of developing symptomatic gallstone disease following bariatric surgery.

DETAILED DESCRIPTION:
To study the incidence and predictors of developing symptomatic gallstone disease following bariatric surgery.

A retrospective study with prospective collective data will be conducted including all patients underwent bariatric surgery in general surgical department, Sohag University between January 2015 and December 2022 who did not have gallstones in the preoperative abdominal ultrasound examinations.

Medical records will be reviewed. Demographic data such as age, gender, BMI, comorbidities as ( DM, hypertension and hyperlipidemia ) and time elapsed between the surgery to post-surgery US examination. The findings of the US examinations will be collected and analyzed. Data will be analyzed to obtain descriptive and inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients underwent bariatric surgery with minimum postoperative follow up period of one year duration will be included in the study.

Exclusion Criteria:

* Patients who had cholecystectomy during the bariatric surgery.
* Pediatric age.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent Bariatric Surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients who develop gall bladder stones after bariatric surgery | one year
  Evalution of gall bladder stone formation postoperaive and its relation with comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No